CLINICAL TRIAL: NCT04060433
Title: Implementation and Evaluation of a Standardized Protocol for Treatment of Restrictive Eating Disorders With Pronounced Starvation During the First Month in Child Psychiatric Outpatient Care. The ROCKETLAUNCH Project
Brief Title: Implementation of Evidence-Based Treatment of Restrictive Eating Disorder With Pronounced Starvation
Acronym: ROCKETLAUNCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lund University Hospital (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Ulf Wallin, MD, PhD Head of Research and Development, Lund University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2019-01852
Record Dates: First submitted 2019-08-12; First posted 2019-08-19 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Anorexia Nervosa; Anorexia Nervosa, Atypical; Avoidant/Restrictive Food Intake Disorder; Starvation
Keywords: Family Therapy; Health Plan Implementation; Outpatients
MeSH Terms: conditions — Anorexia Nervosa; Avoidant Restrictive Food Intake Disorder; Starvation | interventions — Family Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ROCKETLAUNCH project (Experimental): Intensive treatment program with focusing on the implementation of evidence based family therapy
  Interventions: Behavioral: Family Therapy

INTERVENTIONS:
Behavioral: Family Therapy — Swedish version of the evidence based manualized Family Therapy

SUMMARY:
In the Region Skåne in Sweden, the investigators have developed guidelines for providing intensive and evidence-based treatment during the first month in case of severe restrictive eating disorder with pronounced starvation.

The project is aiming at implementing this treatment program in the general Child Psychiatric clinic, with its main focus on the implementation of evidence based family therapy. The study aims to evaluate the implementation of a standardized treatment model during the first month. The outcome will be compared with the patients and families who have been in treatment before the ROCKETLAUNCH project started.

DETAILED DESCRIPTION:
Anorexia nervosa and other restrictive eating disorders with pronounced starvation is one of the most acute and life-threatening conditions in child psychiatry and requires immediate treatment. Anorexia nervosa is the eating disorder which most often causes pronounced starvation, and also has the highest mortality in psychiatry. These conditions are hard to treat, and there are not many successful treatment methods. Family therapy, and more specific family based treatment has so far proved to be the most successful treatment method for the young patient with anorexia nervosa.

For patients presenting with severe underweight, it is critically important to treat starvation and achieve medical stabilization and weight gain as the first priority. Research shows that weight gain during the first month of treatment produces a better outcome. Family-based treatment has the best evidence support to achieve early weight gain for adolescents with anorexia nervosa.

In child and adolescent psychiatry in the Region Skåne in Sweden, a working group have developed guidelines for providing intensive and evidence-based treatment during the first month in case of severe restrictive eating disorder with pronounced starvation.

Whenever a young person diagnosed with an eating disorder is suspected to suffer from starvation, an assessment shall be offered promptly, normally at the latest within fourteen days. If significant cardiac symptoms are reported, assessment must be made within a few days. The treating service should be prepared to offer at least 1-2 visits a week directly at treatment start.

The high-intensity treatment focuses on medical stabilization and weight gain from the first visit. The goal of the treatment during the first month is weight gain of at least 2 kg (exception made for atypical anorexia nervosa with a normal or high weight - where the goal is to achieve medical stabilization). The focus is on helping the patient to conquer starvation. Interventions for normalizing eating will continue after this period.

The project is aiming at implementing this treatment program in the general child psychiatric clinic, with its main focus on the implementation of evidence based family therapy. In the project the investigators have developed two treatment manuals, one for the general family treatment during the first month and one for the family meal.

12 child psychiatric outpatient clinics in the south of Sweden will take part. The study aims to evaluate the implementation of a standardized treatment model during the first month.

The ROCKETLAUNCH project will be running for three years. The study will gather data at three time points.

1. At treatment start
2. After one month
3. At one year follow-up.

The investigators are going to evaluate:

1. The implementation, how the clinical organization and the therapists follow the treatment protocol.
2. The waiting time and the frequency of treatment sessions.
3. Amount of in-patient care.
4. The outcome of the patient, with focus on weight gain and medical stabilization. The investigators will also look at psychological improvement, and evaluate the improvement in specific eating disorders psychopathology and improvement in general psychiatric psychopathology.
5. The health economic cost. The main outcome variables, such as weight gain, waiting time, frequency of treatment sessions and amount of inpatient care will be compared with the patients and families who have been in treatment before the ROCKETLAUNCH project started.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from one in three restrictive Eating Disorders according to DSM-5 criteria: Anorexia Nervosa, Atypical Anorexia Nervosa or Avoidant/Restrictive Food Intake Disorder
* Patient with pronounced starvation
* Patient aged between 7 and 17
* Patient and his/her parents who accept to participate to the study
* Patient comes to treatment for the first time.

Exclusion Criteria:

* Patient who is diagnosed with: psychosis, mental deficiency, organic cerebral disorder, any pathology that interfere with feeding or its regurgitation
* Patient who does not speak Swedish
* Patient who is already in family therapy for an other condition

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-01-20 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 1 month and 12 months
  Change from baseline Body Mass Index (weight in kg/height in m²) at 1 month and 12 months
Medical stabilization | 1 month
  Rate of particapants that have normalized pulse rate and blood pressure.

SECONDARY OUTCOMES:
In-patient treatment | 1 month and 12 months
  Amount of days the patient needs to be hospitalized due to somatic danger
Change from baseline nature and seriousness of eating-disorder symptoms at 1 months and 12 months | 1 month and 12 months
  Patients will complete EDE-Q (Eating Disorder Examination - questionnaire) at baseline, after 1 month and after 12 months. A self-assessment form for eating disorder symptoms.
Change from baseline patient's emotional symptoms at 1 month and 12 months | 1 month and 12 months
  Patients will complete RCADS (Revised Child Anxiety and Depression Scales) at baseline, after 1 month and after 12 months. The RCADS is a 47-item self-report questionnaire, with scales corresponding to separation anxiety disorder (SAD), social phobia (SP), generalized anxiety disorder (GAD), panic disorder (PD), obsessive compulsive disorder (OCD), and major depressive disorder (MDD). The RCADS requires respondents to rate how often each item applies to them. Items are scored 0-3 corresponding to ''never,'' ''sometimes,'' ''often,'' and ''always.'' Higher values represent a worse outcome.

OTHER OUTCOMES:
Therapists treatment fidelity | 1 month
  Percentage of therapists in the study that follow the Swedish Family Therapy for Eating Disorders treatment manual. This will be measured with a questionnaire constructed from the treatment manual and will capture the essential treatment interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf G Wallin, MD PhD, Principal Investigator — Head of Research and Development
Locations (1):
- Psychiatry Skane, Lund University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallin U, Saha S. Implementation of Key Components of Evidence-Based Family Therapy for Eating Disorders in Child and Adolescent Psychiatric Outpatient Care. Front Psychiatry. 2020 Feb 20;11:59. doi: 10.3389/fpsyt.2020.00059. eCollection 2020. PMID 32153439

DOCUMENTS (1):
  • Study Protocol (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT04060433/Prot_000.pdf